### Official Title: <u>Genomic medicine Risk Assessment Care for Everyone (GRACE)</u>

**NCT:** NCT06278883

**IRB Document Date:** 4/26/24

Study ID:IRB202300893 Date Approved: 4/26/2024





# INFORMED CONSENT FORM to Participate in Research, and AUTHORIZATION to Collect, Use, and Disclose Protected Health Information (PHI)

| INTRODUCTION |
|---|
| Name of person seeking your consent: |
| Place of employment & position: |
| GENERAL INFORMATION ABOUT THIS STUDY |
| 1. Name of Participant ("Study Subject") |
| 2. What is the title of this research study (this "Research Study")? |
| GRACE ( <u>G</u> enomic medicine <u>R</u> isk <u>A</u> ssessment <u>C</u> are for <u>E</u> veryone) |
| 3. Whom do you call if you have questions about this Research Study (the "Study Team")? |
| Principal Investigators: |
| Alexander Parker, PhD, MS |

Alexander Parker, PhD, MS
Senior Associate Dean, Research
Director, Precision Medicine
Professor of Epidemiology and Urology
College of Medicine – Jacksonville
University of Florida
904-244-9478
Alexander.Parker@ufl.jax.edu

Lori Orlando, MD Director, Precision Medicine Program Professor of Medicine Duke University

Other research staff:

IRB project: IRB202300893 IRB version: 02/02/2022 PI version: 4/26/2024



Kathryn Carpenter, MS Clinical Research Manager Office of Research Affairs University of Florida-Jacksonville 904-244-5352

#### 4. Who is paying for this Research Study?

The sponsor of this study is the National Institutes of Health (NIH).

#### 5. In general, what do you need to know about this Research Study?

Agreeing to become involved in any research is always voluntary. By signing this form, you are not waiving any of your legal rights. If you decide not to participate in this research, you will not be penalized in any way and you will not lose any benefits to which you are entitled. If you have questions about your rights as a research subject, please call the University of Florida Institutional Review Board (IRB) office at (352) 273-9600.

#### a) In general, what is the purpose of the research? How long will you be involved?

The primary <u>purpose</u> of this study is to help determine the best way to:

- 1. Use family health history information collected by a platform called "MeTree" to understand your personal risk for developing different medical conditions (including certain cancers, heart diseases and/or liver diseases).
- Provide access to genetic counseling and genetic testing for those whose family health history
  information suggests they may have a genetic change that increases their risk for developing
  certain medical conditions (including certain cancers, heart diseases and/or liver diseases). The
  research is focused on ways to help individuals who do not typically have access to these
  resources.

## b) What is involved with your participation, and what are the procedures to be followed in the research?

In this research study you will complete several surveys, enter your family history in a software platform, and receive recommendations about your level of risk for 45 different conditions, in addition to what to discuss with your provider about that risk. There are several possible options for managing risk and one of those may be genetic testing for a hereditary condition. If you receive a recommendation for genetic testing we will provide genetic testing through the study and help you understand what your test results mean.

#### c) What are the likely risks or discomforts to you?

• This research presents minimal risks to you. However, as with all research studies there are potential risks. Potential risks include discomfort and/or distress when you receive your family health history risk and/or genetic test results.

IRB project: IRB202300893 Page **2** of **13** IRB version: 02/02/2022

PI version: 4/26/2024



- There is a very small risk of receiving incorrect genetic results that lead to care that is not needed or to you not receiving care that is needed. This risk is the same if you were to get genetic testing outside of the study.
- If for some reason, we are not able to use your saliva for genetic testing, and you agree to have blood drawn from your arm for genetic testing, you may experience momentary discomfort and/or bruising. Infection, excess bleeding, clotting, or fainting are also possible, although unlikely.
- There is also the potential for loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.
- Fortunately, there is a Federal law called the Genetic Information Nondiscrimination Act (GINA).
   This law makes it illegal for health insurance companies, group health plans, and most employers of over 15 people to discriminate against you based on your genetic information.
   However, it does not protect you against discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.
- GINA does not protect you against discrimination based on an already-diagnosed genetic condition or disease and does not apply to members of the military.
- Some of the questions we will ask you as part of this study may make you feel uncomfortable. You may refuse to answer any of the questions and you may take a break at any time during the study. You may stop your participation in this study at any time.

#### d) What are the likely benefits to you or to others from the research?

You will benefit from taking part in this study because the study will evaluate your risk for 45 different medical conditions including certain cancers, heart diseases and liver diseases. This risk assessment is based on current expert clinical guidelines. If you do have an increased risk you will also be informed about the level of risk and what you can do about it. In addition, if you have genetic testing you might discover a genetic risk for certain cancers, heart diseases, or liver diseases that runs in your family that you did not know about previously. With these pieces of information, you and your healthcare provider may be able to make better decisions about preventive care, and how to keep you healthy.

## e) What are the appropriate alternative procedures or courses of treatment, if any, that might be helpful to you?

Regardless of whether MeTree recommends genetic testing as part of this study, or not, you can discuss genetic testing with your primary care physician and request to have it performed. If you do so, the cost of the testing would be paid by you or your insurance company as part of your care outside this study.

Additional and more detailed information is provided within the remainder of this Informed Consent form. Please read before deciding if you wish to participate in this study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.




#### WHAT CAN YOU EXPECT IF YOU PARTICIPATE IN THIS STUDY?

#### 6. What will be done as part of your normal clinical care?

All appropriate, guideline approved follow-up care based on the results of your familial risk will be done. You may be referred to specialty clinics based on the results of your risk screening and/or genetic testing as part of this study. If you are referred for follow up specialty care, those costs <u>would not</u> be covered by the research study. Your provider may still recommend risk-based screening and testing as part of your routine care even if you don't participate in the study.

#### 7. What will be done only because you are in this Research Study?

If you agree to participate, you will first be asked to complete a baseline survey and enter your family health history (FHH) into an online platform called MeTree. After you complete entering the information in to MeTree, you and your provider will have access to a risk assessment report indicating if you are at increased risk for any conditions and what to talk with your provider about. In addition, you will be asked to complete a survey about the experience of using MeTree.

- We estimate that completing the baseline questionnaire and entering the information requested by MeTree takes on average about 35 minutes to complete.
- We estimate that completing the survey about the MeTree experience will take 8 minutes.

Depending upon the results of the baseline survey and your risk assessment report you may go down one of three pathways:

- 1. If your report indicates you are not at increased risk for any conditions, then 2 weeks later you will be asked to complete a survey about your experience with participating in the study. At this point you will be done with the study.
- 2. If your report indicates that you have a small increase in risk for some conditions (called 'familial' risk) then your report will provide information about steps you can take to manage that risk. Your provider will also have a copy of your report. 2 weeks later you will be asked to complete a survey about your experience with participating in the study. At this point you will be done with the study.
- 3. If your report indicates that you have genetic (inherited) risk for any conditions (called 'hereditary' risk) then you will be recommended to undergo genetic counseling and testing. In the majority of cases, you will learn more about genetic testing from an online genetic information assistant called GIA. You will be sent a video describing GIA and then a link to GIA. If you would like counseling from a person instead you will be able to request that option. You may also decline counseling if you prefer.
  - If you decline counseling then two weeks later, you will be asked to complete a survey about your experience with participating in the study and then your involvement in the study will end.
  - If you undergo counseling and agree to genetic testing then you will be mailed a free saliva test kit with pre-paid return envelope. After collecting your sample in the kit you




will mail it our study partner Invitae (a genetic testing company). If for any reason the test can't be performed on your saliva specimen we can send another kit or have a mobile phlebotomy (blood draw) van meet you at your location of choice to draw blood for the test – at no cost.

- If your genetic test confirms that you do <u>NOT</u> have a change in your DNA ('negative' test result) that increases your risk for an inherited condition then GIA will return those results to you and you will receive a survey 2 weeks later about your experience with participating in the study and then your involvement in the study will end.
- If your genetic test confirms that you <u>DO</u> have a change in your DNA ('positive' test result) that increases your risk for an inherited condition then one of the study genetic counselors will contact you to discuss the results and next steps. Your provider will also be notified of the results. 2 weeks later you will receive a survey about your experience with participating in the study; as well as asking <u>if you would like to share your results with family members</u> so they can receive genetic counseling and testing either through the study or local resources.
  - This is called 'cascade screening' and is important since you share much (but not all)
    of the same genetic code with your family members, so they may also have the
    same genetic risk that you do.
  - The notification of family members is entirely optional. If you decide to provide a list of family members and their contact information on the survey, the study team will: 1) give you a letter you can share with your family members about the test results and how they can get testing, and 2) directly contact them to discuss the result and how to get testing.
- After you complete that survey, you will be finished with the study.

You may withdraw from the study at any point during this process. If you remain in the study, your provider will be provided your risk results and any testing completed.

If any identifiable information was collected as part of this research, it is possible that your research information, with all personally identifiable information removed, could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative. See Addendum on Data Sharing Consent at the end of this form.

If you have any questions now or at any time during this Research Study, please contact one of the Research Team members listed in question 3 of this form.

#### 8. What identifiable health information will be collected about you and how will it be used?

The Research Team will collect the following information for this study:

- Demographic Information, including name and birthdate
- Vital Signs




- Lifestyle Factors
- Medical History
- Family History

The Research Team may collect this information from other healthcare providers, such as laboratories, which are a part of this research. Other professionals at the University of Florida or Shands Hospital who provide study-related care, and the University of Florida Institutional Review Board (IRB), may also collect your health information.

This information will be delivered to the MeTree platform, where you will enter your family health history (FHH) information, which will be housed indefinitely at Duke University on a secured server.

Data that are received by Invitae for saliva and/or blood specimens will be completely de-identified and used to make updates to Invitae's assays, gene classifications, and for other in-house purposes. However, data are not shared, and do not exit the sphere of the company.

The Research Team listed in question 3 above will use or share your health information as described below to carry out this research study.

#### 9. With whom will this health information be shared?

This health information may be shared with:

- the study sponsor (listed in Question 4 of this form);
- United States governmental agencies which are responsible for overseeing research, such as the Food and Drug Administration, the Department of Health and Human Services, and the Office of Human Research Protections;
- government agencies which are responsible for overseeing public health concerns, such as the Centers for Disease Control and federal, state and local health departments, and
- the IRB that reviewed this Research Study and ensures your rights as a Study Subject are protected.

Otherwise, your identifiable health information will not be shared without your permission unless required by law or a court order. Once your health information is shared with those listed above, it is possible that they could share it without your permission because it would no longer be protected by the federal privacy law.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You have been informed that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or




other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information. That is, if you give written consent for the release of information, we cannot withhold that information and we cannot hold responsibility for how that person may use your information.

The Certificate of Confidentiality does not prevent the researchers from disclosing voluntarily, without your consent, information that would identify you as a participant in the research project under the following circumstances. If we learn about child abuse, elder abuse, or intent to harm yourself or others, we will report that information to appropriate authorities.

#### 10. How long will you be in this Research Study?

How long you will be in this study depends on whether you meet criteria for genetic testing or not. For those who do not undergo genetic counseling and testing we expect the study to last no more than 3 weeks. For those who do it may be 1-3 months.

You can choose to stop participating at any time without penalty or loss of any benefits to which you are entitled.

This Authorization to use and share your health information expires at the end of the study, unless you revoke it (take it back) sooner.

#### 11. How many people are expected to take part in this Research Study?

Approximately 2525 people will take part in this study.

#### WHAT ARE THE RISKS AND BENEFITS OF THIS STUDY AND WHAT ARE YOUR OPTIONS?

#### 12. What are the possible discomforts and risks from taking part in this Research Study?

This research presents minimal risks to you. However, as with all research studies there are potential risks. Potential risks include discomfort and/or distress when you receive your family health history risk and/or genetic test results.

There is a very small risk of receiving incorrect genetic results that lead to care that is not needed or to you not receiving care that is needed. This risk is the same if you were to get genetic testing outside of the study

If for some reason, we are not able to use your saliva for genetic testing, and you agree to have blood drawn from your arm for genetic testing, you may experience momentary discomfort and/or bruising. Infection, excess bleeding, clotting, or fainting are also possible, although unlikely.

There is also the potential for loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

Fortunately, there is a Federal law called the Genetic Information Nondiscrimination Act (GINA). This law makes it illegal for health insurance companies, group health plans, and most employers of over 15 people to discriminate against you based on your genetic information. However, it does not protect you against discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA does not protect you against discrimination based on an already-diagnosed genetic condition or disease and does not apply to members of the military.




Some of the questions we will ask you as part of this study may make you feel uncomfortable. You may refuse to answer any of the questions and you may take a break at any time during the study. You may stop your participation in this study at any time.

This Research Study may also include risks that are unknown at this time.

Please note, participating in more than one research study or project may further increase the risks to you. If you are already enrolled in a research study, please inform one of the Research Team members listed in question 3 of this form or the person reviewing this consent with you before enrolling in this or any other research study or project.

During the study, the Research Team will notify you of new information that may become available and might affect your decision to remain in the study.

The University of Florida is required by law to protect your health information. Your health information will be stored in locked filing cabinets or on computer servers with secure passwords, or encrypted electronic storage devices, as required by University policy. However, there is a slight risk that information about you could be released inappropriately or accidentally. Depending on the type of information, a release could upset or embarrass you, or possibly affect your ability to get insurance or a job.

If you wish to discuss the information above or any discomforts you may experience, please ask questions now or call one of the Research Team members listed in question 3 in this form.

#### 13a. What are the potential benefits to you for taking part in this Research Study?

You could benefit from taking part in this study because the study will evaluate your risk for 45 different medical conditions including certain cancers, heart diseases and liver diseases. This risk assessment is based on current expert clinical guidelines. If you do have an increased risk you will also be informed about the level of risk and what you can do about it. In addition, if you have genetic testing you might discover a genetic risk for certain cancers, heart diseases, or liver diseases that runs in your family that you did not know about previously. With these pieces of information, you and your healthcare provider may be able to make better decisions about preventive care, and how to keep you healthy.

#### 13b. How could others possibly benefit from this Research Study?

We hope that in the future the information learned from this study will benefit other people who may be at risk for these conditions as well with greater access to genetic screening based on obtaining a robust family history. As such, you may get some benefit from knowing you participated in research that could help advance medicine and disease prevention for others.

#### 13c. How could the Research Team members benefit from this Research Study?

In general, presenting research results helps the career of a researcher. Therefore, the Research Team listed in question 3 of this form may benefit if the results of this Research Study are presented at scientific meetings or in scientific journals.

One of the study investigators, Dr. Lori Orlando, is a co-founder of a company called MeTree&You. This company allows individuals, outside of a research study, access to the MeTree family health history platform for their care. The research version of MeTree is being used in this study, since it is the risk assessment




platform the researchers have access to, but the goal of the study is not to evaluate MeTree. In addition, the outcomes and analysis of the study are being performed by an unbiased statistician who does not report to Dr. Orlando. The outcomes of this study to do not have any direct benefit for the company.

#### 14. What other choices do you have if you do not want to be in this study?

Regardless of whether MeTree recommends genetic testing as part of this study, or not, you can discuss genetic testing with your provider and request to have it performed. If you do so, the cost of the testing would be paid by you or your insurance company as part of your care outside this study. You may also refuse to authorize the use of your health information, but if you refuse, you may not be allowed to be in this research study or receive any research-related treatment that is only available in this research study. However, your decision not to sign this Authorization will not affect any other treatment you may be eligible to receive.

#### 15a. Can you withdraw from this study?

You may withdraw your consent and stop participating in this Research Study at any time. If you do withdraw your consent, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. If you decide to withdraw your consent to participate in this Research Study for any reason, please contact the Research Team listed in question 3 of this form. They will tell you how to safely stop your participation.

You can also change your mind and take back this Authorization at any time by sending a written notice to the Research Team listed in question 3 of this form to let them know your decision. If you take back this Authorization, the Research Team may only use and disclose your health information already collected for this research study. No additional health information about you will be collected or disclosed to the Research Team. However, if you take back this Authorization, you may not be able to continue in this study. Please discuss this with a member of the Research Team listed in question #3.

#### 15b. Can the Principal Investigator withdraw you from this Research Study?

You may be withdrawn from this Research Study without your consent for the following reasons:

- If you move out of the state of FL
- If you stop receiving care at UF Health

#### WHAT ARE THE FINANCIAL ISSUES IF YOU PARTICIPATE?

#### 16. If you choose to take part in this Research Study, will it cost you anything?

The Sponsor will pay for all Protocol-required medical services that you receive as part of your participation in this study that are not routine, standard-of-care services. All other medical services will be billed to you or your insurance company. You will be responsible for paying any deductible, coinsurance, co-payments, for those services, and for any non-covered or out-of-network services. Some insurance companies may not cover costs associated with research studies. Please contact your insurance company for additional information.




#### 17. Will you be paid for taking part in this Research Study?

You will be compensated up to \$60 for your completion of this study. You will receive \$30 after completing a survey about your experience with the MeTree platform and an additional \$30 when you complete all study components for your risk group.

Your payment for participation in this research study is handled through the University of Florida's Research Participant Payments (RPP) Program. Your information which will include your name, address, and date of birth is protected. Access to the (RPP) Program site is limited to certain staff with the assigned security role. You will be randomly assigned a specific identification (ID) number to protect your identity.

If you have any problems regarding your payment contact the study coordinator.

#### 18. What if you are injured while in this Research Study?

If you are injured as a direct result of your participation in this study, only the professional services that you receive from any University of Florida Health Science Center healthcare provider will be provided without charge. These healthcare providers include physicians, physician assistants, nurse practitioners, dentists or psychologists. Any other expenses, including Shands hospital expenses, will be billed to you or your insurance provider.

You will be responsible for any deductible, co-insurance, or co-payments. Some insurance companies may not cover costs associated with research studies or research-related injuries. Please contact your insurance company for additional information.

The Principal Investigator will determine whether your injury is related to your participation in this study.

No additional compensation is routinely offered. The Principal Investigator and others involved in this study may be University of Florida employees. As employees of the University, they are protected under state law, which limits financial recovery for negligence.

Please contact the Principal Investigator listed in question 3 of this form if you experience an injury or have questions about any discomforts that you experience while participating in this study.

IRB project: IRB202300893 IRB version: 02/02/2022 PI version: 4/26/2024 Study ID:IRB202300893 Date Approved: 4/26/2024



**SIGNATURES** As an investigator or the investigator's representative, I have explained to the participant the purpose, the procedures, the possible benefits, and the risks of this Research Study; the alternative to being in the study; and how the participant's protected health information will be collected, used, and shared with others: Signature of Person Obtaining Consent and Authorization Date You have been informed about this study's purpose, procedures, possible benefits, and risks; the alternatives to being in the study; and how your protected health information will be collected, used and shared with others. You have received a copy of this form. You have been given the opportunity to ask questions before you sign, and you have been told that you can ask questions at any time. You voluntarily agree to participate in this study. You hereby authorize the collection, use and sharing of your protected health information as described above. By signing this form, you are not waiving any of your legal rights. Signature of Person Consenting and Authorizing Date

IRB project: IRB202300893 IRB version: 02/02/2022

PI version: 4/26/2024



## Addendum: Consent To Collect And Share Your Data For Future Research

As part of the research project GRACE (<u>Genomic medicine Risk Assessment Care for Everyone</u>), with the principal investigators – Dr. Alexander Parker and Dr. Lori Orlando, we are seeking your consent to share your research data.

#### **Reason for Storing Your Data:**

This research study is collecting data from you. We would like to make your data available for other research studies that may be done in the future. The research may be about similar diseases or conditions to this study. However, research could also be about unrelated diseases, conditions, or other types of research. These studies may be done by researchers at this institution or other institutions, including commercial entities. Our goal is to make more research possible. We plan to keep your electronic data indefinitely. Some of the data will be deposited in the Database of Genotype and Phenotype (dbGaP), as required by the National Human Genome Research Institute (NHGRI), or other National Institutes of Health data repositories. The dbGaP is a National Institutes of Health (NIH) sponsored repository charged to archive, curate and distribute information produced by studies investigating the interaction of genotype and phenotype in humans.

Your data may be shared with researchers around the world. However, the decision to share your data is controlled by University of Florida, Duke University, and the dbGaP. To get your data, future researchers must seek approval from University of Florida, Duke University, and the dbGaP.

Any researcher using your shared data must agree not to try to identify you.

Your name and identifying information will be removed from any data you provide before they are shared with other researchers. Researchers cannot easily link your identifying information to the data.

## Do I have an option to allow the sharing of my research data with other researchers in addition to those listed above?

It is your choice whether or not to let researchers share your data for research in the future. If you say "yes," you can change your mind later. If you say "no," you can still fully participate in this study.

If you change your mind and no longer wish to have us store or share your data, you should contact the Research Team listed in question 3 of this form. We will do our best to honor your request and to retrieve any data that have been shared with other researchers. However, there may be times we cannot. For example, if we do not have a way to identify your data we will not be able to retrieve them. In addition, if the data have already been used for new research, the information from that research may still be used.

#### **Benefits to You in Sharing Your Data:**

You will not receive any direct benefit from sharing your data. However, sharing your data may contribute to research that could help others in the future.


Study ID:IRB202300893 Date Approved: 4/26/2024



#### Risks to You in Storing and Sharing Your Data:

We will do our best to protect your data during storage and when they are shared. However, there remains a possibility that someone could identify you. There is also the possibility that unauthorized people might access your data. In either case, we cannot reduce the risk to zero.

| Do You Agree to Have Your Research Data Shared for Future Research? |
|---------------------------------------------------------------------|
| Please initial next to your choice: |
| YES, share my data with other research studies in the future. |
| NO, do NOT share my data with other research studies in the future. |
